CLINICAL TRIAL: NCT05035381
Title: Phase II Clinical Study on Efficacy and Safety of PD-1 Inhibitor Combined With Bevacizumab and FOLFIRI Regimen in the Second-line Treatment of Unresectable Recurrent or Metastatic MSI-H Colorectal Cancer
Brief Title: PD-1 Inhibitor Combined With Bevacizumab and FOLFIRI Regimen in the Second-line Treatment of Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJMUCH-GI-CRC02
Record Dates: First submitted 2021-06-21; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-06

CONDITIONS: MSI-H Advanced Colorectal Cancer
MeSH Terms: interventions — pembrolizumab; Immune Checkpoint Inhibitors; Bevacizumab; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experiment Group (Experimental)
  Interventions: Drug: Pembrolizumab (PD-1 Inhibitor) Combined With Bevacizumab and FOLFIRI Regimen

INTERVENTIONS:
Drug: Pembrolizumab (PD-1 Inhibitor) Combined With Bevacizumab and FOLFIRI Regimen — MSI-H colorectal cancer, recurrence and metastasis within 1 year after surgery, or failure of first-line oxaliplatin and fluorouracil chemotherapy for advanced colorectal cancer, PD-1 inhibitors combined with bevacizumab and FOLFIRI regimen
  Other Names: Bevacizumab; Irinotecan; Fluorouracil; Leucovorin

SUMMARY:
MSI-H is a biomarker for solid tumors benefiting from immunotherapy. Recent clinical studies have confirmed that PD-1 inhibitors have a good effect on MSI-H advanced colorectal cancer for first- or second-line treatment. The overall effective rate is 30% to 40%. However, about 30% of patients are resistant to PD-1 inhibitors. Whether PD-1 inhibitors and existing chemotherapeutics and anti-vascular drugs have synergistic effects is worth studying. This study is a phase II prospective clinical study of PD-1 inhibitor combined with bevacizumab and FOLFIRI regimen in the second-line treatment of unresectable recurrent or metastatic MSI-H colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Recurrent or metastatic unresectable colorectal adenocarcinoma confirmed by histology and/or cytology; 2. First-line oxaliplatin-containing chemotherapy has disease progression during chemotherapy or within 6 months after chemotherapy; 3. MSI-H patients confirmed by pathology, MSH2(-) or MSH6(-), for MLH1(-) or PMS2(-) patients need PCR confirmation; 4. According to the RECIST 1.1 standard, there is at least one measurable lesion； 5. Sufficient bone marrow function, liver and kidney function； 6. age greater than 18 years old， less than or equal to 75 years old； 7. ECOG score 0 or 1; expected survival time greater than 3 months; signed informed consent.

Exclusion Criteria:

* 1. For patients who have been treated with PD-1 in the first-line treatment, bevacizumab is allowed in the first-line treatment; 2. Other malignant tumors have been diagnosed within 5 years before the first use of the study drug, except for effectively treated skin basal cell carcinoma, skin squamous cell carcinoma, and/or effectively resected in situ cervical cancer and/or breast cancer; 3. Suffer from any active autoimmune disease or have a history of autoimmune disease; 4. Are suffering from an active infection that requires systemic treatment; 5. The HIV test result is positive; 6. Known to be allergic to certain components of the research drug or similar drugs; 7. Use clinical investigational drugs within 4 weeks before the start of study administration; 8. Major surgery has been performed within 4 weeks before the start of the study administration and has not fully recovered; 9. The patient has a bleeding disorder, and the investigator judges that there is a risk of hemorrhage; 10. Uncontrolled cardiac clinical symptoms or disease heart function, such as severe arrhythmia, uncontrollable hypertension; 11. According to the judgment of the investigator, the subject has other factors that may cause him to be forced to suspend the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to one year

SECONDARY OUTCOMES:
Disease Control Rate | Up to 2 years
Progression-free survival | up to 2 years
Overall survival | up to 3 years
Adverse Events | up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No